CLINICAL TRIAL: NCT05708469
Title: Maternal and Fetal Outcomes of Sugammadex Administration During Pregnancy: A Retrospective Cohort Study
Brief Title: Sugammadex Administration in Pregnancy
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Other Study IDs: sakarya ali eman 001
Record Dates: First submitted 2022-12-22; First posted 2023-02-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sugammadex, Pregnant, Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators aimed to evaluate the maternal and fetal effect of sugammadex in pregnant patients undergoing a non-obstetric surgery. The investigators mainly focused on the short- and long-term adverse effects such as an abortion or a teratogenic effect and that may occur in fetus and the adverse effects that may be seen in mother.

DETAILED DESCRIPTION:
Since the approval in Europe in 2008, sugammadex has been widely studied among pregnant patients in the context of cesarean deliveries. However, the use of sugammadex in pregnant patients undergoing a non-obstetric surgery is not clearly defined. The package insert indicates that there are no data on its use in pregnant women regarding the drug-associated risks. There are some questions raised, and answers needed from the scientific community about the maternal and fetal effect of sugammadex administered in pregnant patients.

This is a retrospective case-control cohort study which was conducted in a single-center territory university hospital. The investigators used the hospital information management system for determining the patients that are eligible for inclusion. Patients operated between January 2017 and june 2022 were included in the study. Patient data was obtained by manual review of anesthesia charts of eligible patients. Pregnant patients who underwent a non-pregnancy surgical intervention within the study period were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were operated under general anesthesia during pregnancy and who used sugammadex during the awakening phase.

Exclusion Criteria:

* Patients with severe hepatic and renal impairment
* Patients with missing data
* Patients with fetal anomaly detected before the procedure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who were operated under general anesthesia during pregnancy and used sugammadex during the recovery period will be included in the study. The study was planned retrospectively. We determined the age group as 18-45.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Fetal outcome | one week postoperatively
  Determined by using APGAR score.
Preterm labor | Labor that starts before 37 completed weeks of pregnancy
  Labor that starts before 37 completed weeks of pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Training and Research Hospital, Serdivan, Sakarya, Turkey (Türkiye)

REFERENCES:
- [Background] Varela N, Lobato F. Sugammadex and pregnancy, is it safe? J Clin Anesth. 2015 Mar;27(2):183-4. doi: 10.1016/j.jclinane.2014.11.015. Epub 2014 Dec 13. No abstract available. PMID 25516396
- [Background] Richardson MG, Raymond BL. Sugammadex Administration in Pregnant Women and in Women of Reproductive Potential: A Narrative Review. Anesth Analg. 2020 Jun;130(6):1628-1637. doi: 10.1213/ANE.0000000000004305. PMID 31283616
- [Background] Torres SM, Duarte DF, Gloria AS, Reis C, Moreira JF, Cunha S, Gomes LL, Dahlem C. Sugammadex administration in pregnant patients undergoing non-obstetric surgery: a case series. Braz J Anesthesiol. 2022 Jul-Aug;72(4):525-528. doi: 10.1016/j.bjane.2021.07.034. Epub 2021 Aug 16. PMID 34411637